CLINICAL TRIAL: NCT00271856
Title: Mindfulness-Based Stress Reduction (MBSR), Stress Arousal and Immune Response in Early HIV
Brief Title: Staying Well: A Clinical Trial of Mindfulness-Based Stress Reduction and Education Groups for HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01AT002024 (NIH); P01AT002024 (NIH)
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: HIV
Keywords: HIV; Meditation; Stress; Randomized Controlled Trial; Complementary Therapies; MBSR; Not on ART medications
MeSH Terms: interventions — Mindfulness-Based Stress Reduction; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0 (Experimental): Mindfulness Based Stress Reduction (MBSR)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- 1 (Active Comparator): HIV education/self-management workshop
  Interventions: Behavioral: HIV-education and self-management workshop

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — 8 week MBSR course
  Other Names: Mindfulness meditation
  Arms: 0
Behavioral: HIV-education and self-management workshop — 8-week group covering a variety of educational topics about managing HIV infection.
  Arms: 1

SUMMARY:
To examine the effects of Mindfulness-Based Stress Reduction (MBSR) and education groups on HIV (Human Immunodeficiency Syndrome) infection. Key outcomes include CD4 and viral load, stress hormones, depression and quality of life.

DETAILED DESCRIPTION:
Stress and depression are associated with more rapid loss of CD4 cells in HIV infection. Interventions that slow the advance of HIV infection and delay the introduction of antiretroviral therapy (ART) could make an important contribution to HIV management in both the developed and developing world. We are conducting a 330 person randomized, controlled clinical trial of MBSR for persons with HIV-1 infection and CD4 T-lymphocyte counts > 250 cells/µm who are not on antiretroviral therapy. Participants are randomized in a 1:1 distribution to either the MBSR intervention or to an education group that will control for the attention and social interaction aspects of MBSR. Participants are evaluated at 0, 3, 6 and 12 months. Key outcome measures at 12 months include differences in CD4 T cell counts, HIV viral load, perceived stress, depression, and positive affect. We are also examining whether MBSR is associated with changes in neuroendocrine function (autonomic nervous system activity, cortisol secretion) and alterations in immune function that may serve as intermediate steps between the neuroendocrine effects of MBSR and CD4 T cell counts, such as changes in T cell activation. A subset of 90 participants will be studied in additional detail using a structured laboratory stress challenge.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Viral Load>100
* CD4 T-Cells>250
* Not on Antiretroviral therapy (ART)
* Ability to Speak English
* Stable address/living situation

Exclusion Criteria:

* Inability to provide informed consent
* Use of ART within the past 120 days
* Any substance abuse,mental health or medical condition that the opinion of the Principal Investigator (PI) would make it difficult for the potential participant to participate in the intervention
* Plans to start ART in the next 12 months
* Previous MBSR training and/or current practice
* Current use or use in past 6 months (mos.) of chemotherapy or immunomodulator drugs, including oral steroids or plans to start in the next 12 mos.
* Initiation of new class of psychiatric medication in past 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Hecht, M.D., Principal Investigator — University of California, San Francisco; Susan Folkman, PhD, Study Director — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2005 to August 2008 through newspaper advertisements, electronic bulletin boards, community postings and fliers in clinics.
Pre-assignment Details: Enrolled participants were screened to determine if inclusion criteria were met. This process included structured phone interviews, medical history review, and laboratory results.
Groups:
- 0 Mindfulness-Based Stress Reduction (MBSR): Mindfulness Based Stress Reduction (MBSR): 8 weekly evening meetings plus one all-day class.
- 1-HIV Education/Self-management: HIV education/self-management workshop: 8 weekly classes.
Period: Overall Study
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Started | 89 | 88
Completed | 78 | 70
Not Completed | 11 | 18
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 87 | 176
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.36) | 40.5 (9.5) | 40.8 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 85 | 86 | 171
Region of Enrollment [Number; unit: participants]
  United States | 89 | 88 | 177

OUTCOME MEASURES:

1. Secondary Outcome: Quality of Life (Short Form Health Survey; SF-36); Cortisol (Basal a.m. and Diurnal Change); T-cell Activation (i.e. CD38-cell Surface Marker) and NK Cell Number and Function; Autonomic Nervous System Activity ; Cell Aging
Time Frame: 3, 6, and 12 months
Reporting Status: Not Posted

2. Primary Outcome: Change in CD4 T-cell Count
Time Frame: baseline to 12 months
Population: Intent to treat (ITT) analyses. Multiple imputation method used for those who started antiretroviral therapy (ART) between 0 and 12 months.
Measure: Mean (95% Confidence Interval); unit: cells/µl
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
cells/µl | -57.1 [-91.2 to -23.0] | -70.3 [-105.5 to -35.1]

3. Primary Outcome: Change in Depression as Measured by Beck Depression Inventory (BDI)
Description: The BDI is a widely used outcome measure for studies of depression. The BDI consists of 21 items that are rated on a 4-point scale according to how severely they are experienced. Scores range from 0-63, with higher scores reflecting greater depression.
Time Frame: baseline to 12 months
Population: ITT analyses.
Measure: Mean (95% Confidence Interval); unit: scores on the scale
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
scores on the scale | -1.85 [-3.66 to -0.035] | -1.68 [-3.48 to 0.13]

4. Primary Outcome: Change in Perceived Stress as Measured by Perceived Stress Scale (PSS)
Description: Perception of stress was measured with the 10-item version of the Perceived Stress Scale. This widely used measure of perceived stress was designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. Participants rate how often they felt or thought a certain way over the past month on a 4-point scale (0 = Never, 4 = Very Often). Scores range from 0-40, with higher scores reflecting greater perceived stress.
Time Frame: baseline to 12 months
Population: ITT analyses.
Measure: Mean (95% Confidence Interval); unit: scores on the scale
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
scores on the scale | -0.58 [-2.14 to 0.99] | -2.03 [-3.35 to -0.71]

5. Primary Outcome: Change in Positive and Negative Affect (PANAS) Positive Affect (PA) Score
Description: Emotion was assessed with the Positive and Negative Affect Schedule (PANAS). The PANAS measures intensity of positive and negative emotions over the past week. The scale consists of 20 items--10 positive and 10 negative emotions. Respondents are asked to indicate how strongly they felt each emotion on a scale from 0 to 4 (not at all to extremely). The Positive Affect (PA) score is derived from summing the scores on the 10 positive emotions. Scores on the PA subscale range from 0-40, with higher scores reflecting more positive affect over the past week.
Time Frame: baseline to 12 months
Population: ITT analyses
Measure: Mean (95% Confidence Interval); unit: scores on the scale
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
scores on the scale | 1.20 [-0.74 to 3.13] | 1.64 [-0.22 to 3.50]

6. Primary Outcome: Change in Positive and Negative Affect Scale (PANAS) Negative Affect (NA) Score
Description: Emotion was assessed with the Positive and Negative Affect Schedule (PANAS). The PANAS measures intensity of positive and negative emotions over the past week. The scale consists of 20 items--10 positive and 10 negative emotions. Respondents are asked to indicate how strongly they felt each emotion on a scale from 0 to 4 (not at all to extremely). The Negative Affect (NA) score is derived from summing the scores on the 10 negative emotions. Scores on the NA subscale range from 0-40, with higher scores reflecting more negative affect over the past week.
Time Frame: baseline to 12 months
Population: ITT analyses.
Measure: Mean (95% Confidence Interval); unit: scores on the scale
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
scores on the scale | -2.17 [-4.25 to -0.085] | -2.63 [-4.27 to -0.99]

7. Primary Outcome: Change in Depression as Measured by the Patient Health Questionnaire-9 (PHQ-9)
Description: We used the Patient Health Questionnaire (PHQ-9) as a measure of depressive symptom severity. The PHQ-9 is the depression module of the self-administered version of the Primary Care Evaluation of Mental Disorders (PRIME-MD) diagnostic instrument. Participants rate the frequency of 9 depression symptoms over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27, with higher scores reflecting greater severity of depressive symptoms.
Time Frame: baseline to 12 months
Population: ITT analyses.
Measure: Mean (95% Confidence Interval); unit: scores on the scale
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Number analyzed (Participants) | 76 | 68
scores on the scale | -1.00 [-2.44 to 0.44] | -1.46 [-2.71 to -0.2]

ADVERSE EVENTS:
Arm/Group | 0 Mindfulness-Based Stress Reduction (MBSR) | 1-HIV Education/Self-management
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/88
Other Adverse Events (participants affected / at risk) | 0/89 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No